CLINICAL TRIAL: NCT06399029
Title: Topical Ruxolitinib as a Treatment of Anti-PD1 Induced Lichenoid Skin Toxicities: a Prospective Single-center Pilot Study
Brief Title: Topical Ruxolitinib Evaluation in Immune-related Lichenoid Skin-Toxicities
Acronym: TRUX-LST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Barbara Meier-Schiesser, Senior physician, Head General Dermatology & Coordinator Skin Cancer Center USZ, Department of Dermatology, University Hospital Zurich, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01779
Record Dates: First submitted 2024-04-25; First posted 2024-05-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Exanthema; Lichenoid Skin Rashes Under Anti-PD1 Tumor Therapy
MeSH Terms: conditions — Exanthema | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Prospective single-center pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Intervention (Experimental): This study will be performed as one-arm with no comparator.
  Interventions: Drug: Ruxolitinib Topical Cream

INTERVENTIONS:
Drug: Ruxolitinib Topical Cream — Ruxolitinib cream will be applied topically twice daily on up to 20% of the body surface over 12 weeks in patients with lichenoid skin toxicity under anti PD1 treatment.
  Other Names: Topical Ruxolitinib (INCB18424)

SUMMARY:
Skin rash during tumor treatment with immunotherapy (anti-PD1 antibody therapy) is a common side effect. If patients suffer from such a skin reaction, they typically suffer from a rash on the chest, back and extremities. The skin reaction is usually treated with cortisone in cream or tablet form. There is already research in humans on the skin reaction under anti-PD1 antibody therapy. Previous studies in humans have shown that certain inflammatory markers are elevated. It is also know that the study drug can help to reduce these inflammatory markers. However, there is currently not enough data available whether the study drug can actually reduce inflammation in the skin in a rash under anti-PD1 antibody therapy. The investigators are therefore examining in this study whether the study drug is effective and well tolerated in a skin rash under anti-PD1 antibody therapy. The study drug contains the active ingredient ruxolitinib and is applied as a cream. The study drug is approved for other skin diseases (vitiligo and atopic eczema) in the USA and in countries of the European Union (EU). Approval in Switzerland is still pending. Only once the efficacy of the study drug against skin rashes under anti-PD1 antibody therapy has been scientifically investigated and proven can it be approved and used as a therapy in Switzerland. In this study, the participants are not divided into groups. Each study patient receives the test substance.

ELIGIBILITY:
Inclusion Criteria:

Adult patients eligible for this inclusion in this study have to fulfil all the following criteria:

* Indication: lichenoid skin toxicities / rash which has developed under / after anti-PD-1 therapy.
* Male and Female patients ≥18 years of age
* Patients that are able to speak and read German or English.
* The subject was informed and gave his/her consent to the Institutional Review Boards (IRB)/Independent Ethics Committee (IEC) -approved informed consent

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for the inclusion in this study:

* Patient suffering other skin disease resembling lichenoid skin lesions under anti-PD-1 therapy.
* Acute psychiatric illness or acute crisis.
* Contraindications to ruxolitinib, e.g. known hypersensitivity or allergy
* Topical glucocorticosteroids, topical calcineurin inhibitors and UV light therapy are not allowed during the study or for 1 week before the study beginning. Other JAK inhibitors or potent immunosuppressants such as azathioprine or cyclosporine are not allowed during the study or for 8 weeks before the study beginning.
* Women who are pregnant or breast feeding *
* Intention to become pregnant during the course of the study
* Known or suspected non-compliance, drug or alcohol abuse.
* Patients with an active, serious infection, including localized infections.
* Inability to follow the procedures of the study due to language problems, psychological disorders, dementia of the participant.
* Participation in another study with topical or oral ruxolitinib within the 30 days preceding and during the present study.
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

  * Participants must avoid pregnancy during the study. A blood pregnancy test is required before start of therapy, with regular urine tests throughout. Lactating individuals are ineligible.

Participants must use effective contraceptives, either:

* An ovulation-inhibiting method (e.g., pill, injectable, implant, patch, or vaginal ring) or
* An intrauterine device (IUD).
* Contraception should extend one week post-study. If pregnancy occurs during or within one week after the study, participants should notify the overseeing physician immediately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving at least 90% improvement of rash at week 12. | week 12
  The improvement of rash is defined on the physician global assessment score (PGA) and on the body surface area (BSA).
  PGA: measures the overall response to treatment as assessed by the physician; scale 0-4
  Reduction of PGA (e.g. PGA 4 to PGA0) will be converted into percentage: decrease of PGA of 1 point on a scale from 0 to 4 shows a decrease of 25%, decrease of 4 points shows a decrease of 100%.
  This value (percentage of PGA decrease) will be combined with the reduction of BSA (percentage) and will result in the improvement of rash.

SECONDARY OUTCOMES:
Proportion of patients achieving 75% improvement of rash at week 12. | week 12
  The improvement of rash is defined on the physician global assessment score (PGA) and on the body surface area (BSA).
  PGA: measures the overall response to treatment as assessed by the physician; scale 0-4
  Reduction of PGA (e.g. PGA 4 to PGA0) will be converted into percentage: decrease of PGA of 1 point on a scale from 0 to 4 shows a decrease of 25%, decrease of 4 points shows a decrease of 100%.
  This value (percentage of PGA decrease) will be combined with the reduction of BSA (percentage) and will result in the improvement of rash.
Proportion of patients achieving 50% improvement of rash at week 12. | week 12
  The improvement of rash is defined on the physician global assessment score (PGA) and on the body surface area (BSA).
  PGA: measures the overall response to treatment as assessed by the physician; scale 0-4
  Reduction of PGA (e.g. PGA 4 to PGA0) will be converted into percentage: decrease of PGA of 1 point on a scale from 0 to 4 shows a decrease of 25%, decrease of 4 points shows a decrease of 100%.
  This value (percentage of PGA decrease) will be combined with the reduction of BSA (percentage) and will result in the improvement of rash.
Percentage change from body surface area at baseline to week 2, 4, 8 and 12 | baseline, week 2, 4, 8 and 12
  Calculation of the affected body surface area as a percentage.
Proportion of patient reported outcome: Itch Numerical Rating Scale (Itch NRS) | baseline, week 2, 4, 8 and 12
  Itch Numerical Rating Scale (Itch NRS): 2 questions, rating the itch intensity on a scale from 0 to 10 points
Proportion of patient reported outcome: Dermatology Life Quality Index (DLQI) | baseline, week 2, 4, 8 and 12
  Dermatology Life Quality Index (DLQI): 10 questions, summing the score of each question resulting in a minimum of 0 and a maximum of 30 points
Proportion of patient reported outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) | baseline, week 2, 4, 8 and 12
  Treatment Satisfaction Questionnaire for Medication (TSQM): The TSQM is a questionnaire used to measure patient satisfaction with medication. The score ranges from 0 to 100 points
Proportion of patient reported outcome: Five Well-Being Index (WHO-5) | baseline, week 2, 4, 8 and 12
  Five Well-Being Index (WHO-5): a short self-reported measure of current mental wellbeing. It consists of five statements, which respondents rate according to a scale between 0 to 5

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Zürich, Department Dermatology, Zurich, Switzerland